CLINICAL TRIAL: NCT02288156
Title: Elaboration of Patient-friendly Treatment Strategy With Capsaicin Nasal Spray in Patients With Idiopathic Rhinitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TBM
Record Dates: First submitted 2014-11-06; First posted 2014-11-11 (Estimated); Results first posted 2021-01-12 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2021-05

CONDITIONS: Non-allergic Rhinitis
MeSH Terms: conditions — Common Cold | interventions — Capsaicin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 0.1mM (Active Comparator)
  Interventions: Drug: Capsaicin
- 0.01mM (Experimental)
  Interventions: Drug: Capsaicin
- 0.001mM (Experimental)
  Interventions: Drug: Capsaicin
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Capsaicin — via nasal spray
  Arms: 0.001mM; 0.01mM; 0.1mM
Drug: placebo — via nasal spray
  Arms: Placebo

SUMMARY:
Chronic rhinitis is affecting more than 200 million people worldwide. Its prevalence is estimated to be as high as 30% of the Western population. Rhinitis is defined as symptomatic inflammation of the inner lining of the nose and is characterized by the following symptoms: rhinorrhea, nasal blockage, nasal itching and/or sneezing. The cut-off point for defining rhinitis as chronic rhinitis is considered to be persisting symptoms for over more than twelve weeks Chronic rhinitis can be divided into three major subgroups; based on the knowledge of the major etiological factor: infectious rhinitis, allergic rhinitis and non-allergic, non-infectious rhinitis, in literature also referred to as nonallergic rhinitis. Non-inferiority in efficacy of the two novel treatment regimes i.e. capsaicin nasal spray 0,01mM (2puffs/nostril/day) during 4 weeks and capsaicin nasal spray 0,001mM (2puffs/nostril/day) during 4 weeks compared to the current treatment of capsaicin nasal spray 0,1mM (5/day administered on a single day) with regard to the change from baseline in VAS for major nasal symptom on week 4.

(Estimated placebo effect is 25%.)

ELIGIBILITY:
Inclusion Criteria:

* idiopathic rhinitis patients with at least 2 persistent (> 12w) rhinological symptoms (nasal discharge, sneezing, nasal congestion) for an average of at least 1 h per day,
* idiopathic rhinitis patients with a total nasal symptoms score (TNS) of 5 or more on a visual analogue scale (VAS).
* Age > 18 and < 65 years.
* Written informed consent.
* Willingness to adhere to visit schedules.
* Adequate contraceptive precautions in female patients with childbearing potential.

Exclusion Criteria:

* Patients with concomitant allergic rhinitis, demonstrated by positive skin prick test (Hal reagents) and/or immunoglobins E in blood. *
* Patients with structural abnormalities: nasal polyps, severe septal deviation (septum reaching concha inferior or lateral nasal wall), septal perforation, hypertrophy of the inferior turbinates.
* Patients with local allergic rhinitis (LAR) or entopy.
* Systemic steroid treatment less than 4 weeks before the inclusion in the study, nasal steroid spray less than 4 weeks before the inclusion, oral leukotriene antagonists or long-acting antihistamines less than 2 weeks before the inclusion.
* Inability of the patient to stop taking medication affecting nasal function like ß-blockers.
* History of prolonged use or abuse of decongestant nasal spray like xylometazoline spray and/or use or abuse of decongestive oral medication.
* Evidence of infectious rhinitis/rhinosinusitis or common cold within 4 weeks prior to inclusion.
* Pregnancy or lactation. **
* Any disorder of which might compromise the ability of a patient to give truly informed consent for participation in this study.
* Enrollment in other investigational drug trial(s) or receiving other investigational agent(s) for any other medical condition.
* Contra-indications for the use of local anesthesia (cocaine 5%).
* Smoking or occupational exposure to irritants (like hypochlorite, persulfates, isocyanates).
* Nasal malignancies or severe comorbidity like granulomatosis or vasculitis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-07; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Hellings, Prof. Dr., Principal Investigator — UZ Leuven
Locations (1):
- ORL, Leuven, Vlaams-Brabant, Belgium

REFERENCES:
- [Derived] Van Gerven L, Steelant B, Cools L, Callebaut I, Backaert W, de Hoon J, Ampe E, Talavera K, Hellings PW. Low-dose capsaicin (0.01 mM) nasal spray is equally effective as the current standard treatment for idiopathic rhinitis: A randomized, double-blind, placebo-controlled trial. J Allergy Clin Immunol. 2021 Jan;147(1):397-400.e4. doi: 10.1016/j.jaci.2020.04.054. Epub 2020 May 19. No abstract available. PMID 32439432

RESULTS

PARTICIPANT FLOW:
Groups:
- 0,1mM; 0,01mM; 0.001mM: Capsaicin: via nasal spray
Period: Overall Study
Arm/Group | 0,1mM | 0,01mM | 0.001mM | Placebo
Started | 20 | 20 | 20 | 20
Completed | 16 | 16 | 18 | 18
Not Completed | 4 | 4 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 0,1mM | 0,01mM | 0.001mM | Placebo | Total
Number analyzed (Participants) | 16 | 16 | 18 | 18 | 68
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50 (14) | 45 (10) | 48 (14) | 45 (15) | 47 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 9 | 10 | 35
  Male | 7 | 9 | 9 | 8 | 33
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Change in Visual Analogue Scale for Major Nasal Symptoms
Description: patients score their main nasal complaints from 0 to 10 on a scale of 10, with 0 meaning no complaints and 10 meaning the worst complaints. This is done at baseline and after 4 weeks of treatment
Time Frame: Baseline and week 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0,1mM | 0,01mM | 0.001mM | Placebo
Number analyzed (Participants) | 16 | 16 | 18 | 18
score on a scale
  Week 4 | 3.66 (2.78) | 4.29 (2.92) | 4.49 (2.93) | 5.6 (1.67)
  Baseline | 8.36 (1.68) | 8.03 (1.36) | 7.74 (1.48) | 8.24 (1.51)

2. Secondary Outcome: Change in Visual Analogue Scale for Individual Nasal Symptoms
Description: patients score all kinds of nasal symptoms from 0 to 10 on a scale of 10, with 0 meaning no complaints and 10 meaning the worst complaints. This is done at baseline and after 4 weeks of treatment
Time Frame: Baseline, week 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.1mM | 0.01mM | 0.001mM | Placebo
Number analyzed (Participants) | 16 | 16 | 18 | 18
score on a scale
  Rhinorrhea Baseline | 7.594 (2.569) | 5.994 (3.305) | 4.212 (3.318) | 5.806 (3.751)
  Rhinorrhea Week 4 | 2.738 (2.796) | 2.313 (2.572) | 2.383 (2.868) | 3.018 (2.325)

3. Secondary Outcome: Therapeutic Response in All Treatment Regimes
Description: Evaluation of the therapeutic response (TRE) on a scale from 1 (= no relief of symptoms) to 5 (= total relief of symptoms).
Time Frame: week 4
Measure: Number; unit: percentage of patients with improvement
Arm/Group | 0.1mM | 0.01mM | 0.001mM | Placebo
Number analyzed (Participants) | 16 | 16 | 18 | 18
percentage of patients with improvement | 70 | 82 | 35 | 23

4. Secondary Outcome: Change of Nasal Hyperreactivity in All Treatment Modalities.
Description: change in the number of participants with nasal hyperreactivity in all treatment modalities
Time Frame: baseline, week 4
Measure: Number; unit: participants
Arm/Group | 0.1mM | 0.01mM | 0.001mM | Placebo
Number analyzed (Participants) | 16 | 16 | 18 | 18
participants
  Baseline | 7 | 9 | 8 | 9
  week 4 | 5 | 5 | 4 | 8

5. Secondary Outcome: Number of Adverse Events in All Treatment Groups
Description: All reported AEs were entered into the AE section so please see AE table for specifics.
Time Frame: week 4
Population: All reported AEs were entered into the AE section so please see AE section for specifics.
Measure: Number; unit: Total number of events
Arm/Group | 0.1mM | 0.01mM | 0.001mM | Placebo
Number analyzed (Participants) | 16 | 16 | 18 | 18
Total number of events | 27 | 24 | 32 | 29

6. Secondary Outcome: Number of Patients Without Improvement of Symptoms at the End of the Trial in All Treatment Modalities
Time Frame: week 4, 12 and 26
Measure: Count of Participants; unit: Participants
Arm/Group | 0.1mM | 0.01mM | 0.001mM | Placebo
Number analyzed (Participants) | 16 | 16 | 18 | 18
Participants | 10 | 6 | 10 | 12

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | 0,1mM | 0,01mM | 0.001mM | Placebo
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16 | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 10/16 | 8/16 | 14/18 | 12/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0,1mM (N=16) | 0,01mM (N=16) | 0.001mM (N=18) | Placebo (N=18)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Eye infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye irritation (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye Pruritus (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eyelid operation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Food poisoning (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Head discomfort (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Influenza (Infections and infestations) | 1 (1) | 1 (1) | 3 (3) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Laryngitis (Infections and infestations) | 1 (1) | 1 (2) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mite allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 1 (1) | 1 (1)
Nasal crusting (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
nasopharyngitis (Infections and infestations) | 7 (11) | 5 (9) | 8 (9) | 6 (9)
oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (2) | 0 (0) | 3 (5) | 2 (2)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Throat clearing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tonsilitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-12-09): https://cdn.clinicaltrials.gov/large-docs/56/NCT02288156/Prot_SAP_001.pdf